CLINICAL TRIAL: NCT07313137
Title: Antiplatelet Use in All-Cause Dementia and Dementia Subtypes Among Older Adults: A Population-Based Cohort Study
Brief Title: Antiplatelet Use in Dementia Subtypes
Status: Completed | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ZEHRA SARIKAYA DEMIRBAS, MD, Geriatrics Fellow, Gulhane Training and Research Hospital
Other Study IDs: GTRH-ANTIPL-DEM-01
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Dementia Disorder
Keywords: Antiplatelet therapy; Older adults; Dementia subtypes
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dementia cohort: This cohort includes older adults aged 65 years and older diagnosed with dementia who were evaluated in a tertiary geriatric outpatient clinic. No intervention was assigned, as this is a retrospective observational study.

SUMMARY:
This population-based retrospective cohort study aimed to evaluate the appropriateness of antiplatelet therapy use among older adults with all-cause dementia and across different dementia subtypes. Medical records of patients aged 65 years and older who were evaluated at a tertiary-level geriatric outpatient clinic were reviewed. Dementia subtypes were classified according to internationally accepted diagnostic criteria. Patterns of antiplatelet use were assessed in accordance with current guideline recommendations. The study sought to determine the appropriateness of antiplatelet use across dementia subtypes and to describe real-world prescribing practices in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older.
* Diagnosis of dementia based on internationally accepted diagnostic criteria.
* Evaluation at a tertiary-level geriatric outpatient clinic.

Exclusion Criteria:

* Patients with incomplete or inaccessible medical records.
* Individuals with missing data on antiplatelet therapy use.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of older adults aged 65 years and older with a diagnosis of dementia who were evaluated in a tertiary-level geriatric outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Appropriateness of antiplatelet therapy use | At baseline (first geriatric outpatient clinic visit)
  Assessment of the appropriateness of antiplatelet therapy use according to current guideline recommendations among older adults with dementia.

IPD SHARING:
Plan to Share IPD: No